CLINICAL TRIAL: NCT03498677
Title: Effects of Question Section Order on Prioritization of Items by Stakeholder Groups in an Online Delphi Study
Brief Title: Protocol Lab for Online Trial Delphi and Question Effects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThinkWell (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PLOT-D Question Effects
Record Dates: First submitted 2018-04-01; First posted 2018-04-17 (Actual); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Behavior, Adaptive; Decision Analysis
Keywords: online trial; decision analysis
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Method of presentation one (Active Comparator)
  Interventions: Behavioral: presentation order
- Method of presentation two (Active Comparator)
  Interventions: Behavioral: alternative presentation order

INTERVENTIONS:
Behavioral: presentation order — section presentation one
  Arms: Method of presentation one
Behavioral: alternative presentation order — section presentation two
  Arms: Method of presentation two

SUMMARY:
This study nested as a randomized controlled trial within an online Delphi and will assess the impact of using different question section groupings to provide aggregate feedback to participants in an online Delphi study.

DETAILED DESCRIPTION:
A similar assessment has been done during the development of a core outcome for critical care trials set with a nested study examining the impact of question order on prioritization of outcomes. Research reports different stakeholders groups may differ in how they value or prioritize research questions and outcomes and it is recommended that each group should be adequately represented.

The Protocol Lab for Online Trials-Delphi (PLOT-D) study will use an online Delphi combined with participatory action research to inform the development of a multi-use protocol template for writing protocols for self-recruited online trials of interventional self-management. The Protocol lab will use the Delphi findings, along with earlier research to redesign a series of protocols for online randomized trials with the aim of providing support for citizens to work alongside researchers to build participatory health trials online.

ELIGIBILITY:
Inclusion Criteria:

* Protocol lab for online trials Delphi (PLOT-D) participants

Exclusion Criteria:

* None if inclusion criteria are met

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 385 (Actual)
Dates: Start 2018-05-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Context effects of question order | Up to 20 weeks or study completion
  measure to what extent question section order changes context response between conditions

SECONDARY OUTCOMES:
Question section presentation order | Up to 20 weeks or study completion
  response differences amongst stakeholder groups randomized to 1 of 2 presentation order conditions
Retention | Up to 20 weeks or study completion
  difference in number of items retained at the end of the first Delphi round by randomized assignment to condition

CONTACTS AND LOCATIONS:
Overall Officials: Amy Price, PhD, Principal Investigator — University of Oxford
Locations (1):
- ThinkWell, Oxford, Oxfordshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Aggregated de-identified data will be available on reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Post-study, five years
Access Criteria: Contact study investigator

REFERENCES:
- [Background] Brookes ST, Chalmers KA, Avery KNL, Coulman K, Blazeby JM; ROMIO study group. Impact of question order on prioritisation of outcomes in the development of a core outcome set: a randomised controlled trial. Trials. 2018 Jan 25;19(1):66. doi: 10.1186/s13063-017-2405-6. PMID 29370827
- [Background] Potter S, Brookes ST, Holcombe C, Ward JA, Blazeby JM. Exploring methods the for selection and integration of stakeholder views in the development of core outcome sets: a case study in reconstructive breast surgery. Trials. 2016 Sep 23;17(1):463. doi: 10.1186/s13063-016-1591-y. PMID 27664072
- [Background] Snow R, Crocker JC, Crowe S. Missed opportunities for impact in patient and carer involvement: a mixed methods case study of research priority setting. Res Involv Engagem. 2015 Aug 4;1:7. doi: 10.1186/s40900-015-0007-6. eCollection 2015. PMID 29062496
- [Background] Sinha IP, Smyth RL, Williamson PR. Using the Delphi technique to determine which outcomes to measure in clinical trials: recommendations for the future based on a systematic review of existing studies. PLoS Med. 2011 Jan 25;8(1):e1000393. doi: 10.1371/journal.pmed.1000393. PMID 21283604
- [Background] Fletcher AJ, Marchildon GP. Using the Delphi Method for Qualitative, Participatory Action Research in Health Leadership. International Journal of Qualitative Methods 2014;13:1-18
- [Background] Brice A, Price A, Burls A. Creating a database of internet-based clinical trials to support a public-led research programme: A descriptive analysis. Digit Health. 2015 Nov 20;1:2055207615617854. doi: 10.1177/2055207615617854. eCollection 2015 Jan-Dec. PMID 29942546
- [Background] Bagley HJ, Short H, Harman NL, Hickey HR, Gamble CL, Woolfall K, Young B, Williamson PR. A patient and public involvement (PPI) toolkit for meaningful and flexible involvement in clinical trials - a work in progress. Res Involv Engagem. 2016 Apr 27;2:15. doi: 10.1186/s40900-016-0029-8. eCollection 2016. PMID 29062516
- [Background] Price A, Albarqouni L, Kirkpatrick J, Clarke M, Liew SM, Roberts N, Burls A. Patient and public involvement in the design of clinical trials: An overview of systematic reviews. J Eval Clin Pract. 2018 Feb;24(1):240-253. doi: 10.1111/jep.12805. Epub 2017 Oct 27. PMID 29076631
- [Background] Altman DG. Practical statistics for medical research. London: Chapman and Hall; 1991